CLINICAL TRIAL: NCT00879606
Title: Efficacy and Safety Evaluation of ALT-836 in Patients With Sepsis and Acute Lung Injury/Acute Respiratory Distress Syndrome
Brief Title: Anti-TF Antibody (ALT-836) to Treat Septic Patients With Acute Lung Injury or Acute Respiratory Distress Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Altor BioScience (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA-ALT-836-01-08; NHLBI/NIH-5R44HL082397-03
Record Dates: First submitted 2009-04-08; First posted 2009-04-10 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-03

CONDITIONS: Sepsis; Acute Lung Injury; Acute Respiratory Distress Syndrome
Keywords: Sepsis; Acute Lung Injury; Acute Respiratory Distress Syndrome; ALI/ARDS; Lung Disease
MeSH Terms: conditions — Sepsis; Acute Lung Injury; Respiratory Distress Syndrome; Lung Diseases | interventions — ALT-836

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will be randomized to receive ALT-836.
  Interventions: Drug: ALT-836
- 2 (Placebo Comparator): Patients will be randomized to receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALT-836 — In the first part of this study, recombinant chimeric anti-tissue factor antibody ALT-836 was administered as a single dose (0.06 mg/Kg) via intravenous infusion over 15 minutes. In the second part of this study, up to four doses (0.06 mg/Kg) of ALT-836 will be administered via intravenous infusion over 15 minutes.
  Other Names: Formerly TNX-832; Sunol-cH36
  Arms: 1
Drug: Placebo — In the first part of this study, a single dose of Placebo was administered via intravenous infusion over 15 minutes. In the second part of this study, up to four doses of Placebo will be administered via intravenous infusion over 15 minutes.
  Arms: 2

SUMMARY:
This is a prospective, randomized (1:1), double-blind, multi-center, Phase II clinical study to test the safety and efficacy of a recombinant chimeric anti-tissue factor antibody (ALT-836) versus placebo in patients with sepsis and acute lung injury/acute respiratory distress syndrome (ALI/ARDS). This study was divided into two parts and the first part of the study has been completed. In the first part of the study, sixty patients were randomized at a 1:1 ratio to receive one dose of the study drug or placebo. In the second part of the study, ninety patients will be randomized at a 1:1 ratio to receive a multi-dose treatment regimen of single doses every 72 hours up to a maximum of 4 doses of the study drug or placebo, provided there are no safety concerns.

DETAILED DESCRIPTION:
Tissue factor (TF)-dependent procoagulant activity and associated inflammatory processes may play a role in the severity and progression of ALI/ARDS. Recent studies demonstrated that TF levels were elevated in plasma and pulmonary edema fluid of ARDS/ALI patients compared to control patients with hydrostatic pulmonary edema. These higher plasma TF levels were correlated with increased mortality, fewer ventilation-free days, the presence of disseminated intravascular coagulation and the presence of sepsis in patients with ALI/ARDS, suggesting that systemic activation of coagulation may be clinically important in ALI/ARDS. Moreover, the pulmonary TF levels in patients with ALI/ARDS were found to range between 0.5 and 2 nM, approximately 100-fold higher than simultaneous plasma levels, suggesting an intra-alveolar source of TF. Thus, anti-TF antibody blockage of TF activity may therefore provide an effective therapeutic mechanism for the treatment of inflammatory disorders such as ALI and ARDS. This study will test the hypothesis that administration of anti-TF antibody (ALT-836) to septic patients with ALI/ARDS will improve the clinical outcome by shortening the duration of mechanical ventilation for these patients.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Suspected or proven infection
2. Hypoxemia: PaO2/FiO2is ≤300 mm Hg
3. Bilateral infiltrates consistent with pulmonary edema
4. Positive-pressure mechanical ventilation through an endotracheal tube
5. No clinical evidence of left atrial hypertension to explain bilateral infiltrates
6. Presence of at least three of the four SIRS criteria. If only two criteria are evidenced, one must be temperature or WBC

Criteria 2 and 3 must occur within a 24-hour interval. The 48-hour enrollment time window begins when criteria 2, 3, and 4 are met.

EXCLUSION CRITERIA:

1. <18 years
2. Inability to obtain consent
3. Patient, surrogate, or physician not committed to full support
4. Moribund state in which death was perceived to be imminent
5. Morbid obesity
6. Malignancy or other irreversible disease or condition for which 6-month mortality is estimated to be >50%
7. Known HIV positive with known end stage processes
8. Prior cardiac arrest requiring CPR without fully demonstrated neurological recovery; or New York Heart Association Class IV
9. Pregnant or nursing
10. ALI/ARDS induced by mechanical or chemical injury directly to the lung (including burns, trauma, and near drowning)
11. >48 hours since all inclusion criteria are met
12. Neuromuscular disease that impairs ability to ventilate without assistance
13. Severe chronic respiratory disease, severe pulmonary hypertension, or ventilator dependency
14. Chest wall deformity resulting in severe exercise restriction, secondary polycythemia, or respirator dependent
15. History of organ transplant (including bone marrow)
16. Severe chronic liver disease, as determined by a Child-Pugh Score >10
17. Hemoglobin persistently < 7.0 g/dL
18. Platelet count <50,000/mm3
19. Prolonged INR >3
20. Bleeding disorders unless corrective surgery has been performed
21. Active internal bleeding
22. Major surgery within 24 hours before study drug infusion, or evidence of active bleeding postoperatively, or plan for any major surgery within 3 days after study drug infusion.
23. Diffuse alveolar hemorrhage from vasculitis
24. Known bleeding diathesis
25. Presence of an epidural catheter or lumbar puncture within 48 hours before study drug infusion or anticipation of receiving an epidural catheter or a lumbar puncture within 48 hours after study drug infusion
26. Stroke within 3 months of study entry
27. Trauma with an increased risk of life-threatening bleeding
28. A history of severe head trauma that required hospitalization, or intracranial surgery within two months of study entry
29. Any history of intracerebral arteriovenous malformation, cerebral aneurysm, or central nervous system mass lesion
30. Uses of certain medications or treatment regimens such as chemotherapy, unfractionated heparin, low-molecular-weight heparin, Warfarin, antithrombin III, acetylsalicylic acid, glycoprotein IIb/IIIa antagonists, thrombolytic therapy, and activated Protein C are restricted.
31. Participation in another experimental medication study within 30 days of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-04; Primary Completion 2012-10 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Safety profile of the study drug | Throughout the 28 days following treatment
Number of ventilator-free days at Day 28 | Determined at Day 28

SECONDARY OUTCOMES:
Mortality at Day 7, 14, 21, 28 and 60 | Determined at Day 7, 14, 21, 28 and 60
Length of hospitalization at Day 28 | Determined at Day 28
Length of ICU stay at Day 28 | Determined at Day 28
Number of Non-pulmonary organ failure free days at Day 28 | Determined at Day 28
Changes in physiological variables of lung injury | Throughout the 28 days following treatment
Changes in disease severity and lung injury scores | Throughout the 28 days following treatment
Effects of the study drug and the etiology of the disease (i.e. pulmonary or extra-pulmonary origin) | Determined at Day 28
Pharmacokinetics & Pharmacodynamics | Throughout the 28 days following treatment
Immunogenicity | Throughout the 28 days following treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hing C Wong, PhD, Study Chair — Altor BioScience
Locations (20):
- United States (20):
  - Los Angeles County and USC Medical Center, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - Stanford University, Stanford, California
  - Yale University, New Haven, Connecticut
  - Northwestern University, Chicago, Illinois
  - West Suburban Hospital Medical Center, Oak Park, Illinois
  - Illinois Lung and Critical Care Institute, Peoria, Illinois
  - University of Iowa, Iowa City, Iowa
  - Kentucky Lung Clinic, Hazard, Kentucky
  - University of Louisville-Division of Pulmonary and Critical Care, Louisville, Kentucky
  - Baystate Medical Center, Springfield, Massachusetts
  - Saint Luke's Hospital, Kansas City, Missouri
  - Saint Louis University, St Louis, Missouri
  - Mercy Hospital St. Louis, St Louis, Missouri
  - Mount Sinai Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Piedmont Respiratory Research Foundation, Greensboro, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - University of Oklahoma, Oklahoma City, Oklahoma

REFERENCES:
- [Derived] Morris PE, Steingrub JS, Huang BY, Tang S, Liu PM, Rhode PR, Wong HC. A phase I study evaluating the pharmacokinetics, safety and tolerability of an antibody-based tissue factor antagonist in subjects with acute lung injury or acute respiratory distress syndrome. BMC Pulm Med. 2012 Feb 16;12:5. doi: 10.1186/1471-2466-12-5. PMID 22340260
- See also: Altor Bioscience Corporation, Miramar, Florida, US — http://www.altorbioscience.com